CLINICAL TRIAL: NCT03621956
Title: Cardiac and Cerebral Hemodynamics With Umbilical Cord Milking Compared With Early Cord Clamping: A Randomized Cluster Crossover Trial
Brief Title: Cardiac and Cerebral Hemodynamics With Umbilical Cord Milking Compared With Early Cord Clamping
Acronym: MINVINIRS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sharp HealthCare (Other)
Collaborators: Sharp Mary Birch Hospital for Women & Newborns (Other)
Responsible Party: Principal Investigator, Anup Katheria, M.D., Director, Neonatal Research Institute, Sharp HealthCare
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MINVI_NIRS Sub-study
Record Dates: First submitted 2018-08-06; First posted 2018-08-09 (Actual); Results first posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Birth Asphyxia With Neurologic Involvement
Keywords: Near-Infrared Spectroscopy
MeSH Terms: interventions — Umbilical Cord Clamping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Umbilical Cord Milking (Active Comparator): At delivery, the umbilical cord is grasped, and blood is pushed toward the infant 4 times before the cord is clamped. This procedure infuses a placental transfusion of blood into the infant and can be done in 15-20 seconds.
  Interventions: Procedure: Umbilical Cord Milking
- Early Cord Clamping (Active Comparator): The umbilical cord is clamped within 30 seconds of delivery.
  Interventions: Procedure: Early Cord Clamping

INTERVENTIONS:
Procedure: Umbilical Cord Milking — At delivery, the umbilical cord is grasped, and blood is pushed toward the infant 4 times before the cord is clamped. This procedure infuses a placental transfusion of blood into the infant and can be done in 15-20 seconds.
  Arms: Umbilical Cord Milking
Procedure: Early Cord Clamping — The umbilical cord is clamped within 30 seconds of delivery.
  Arms: Early Cord Clamping

SUMMARY:
3 clinical sites enrolling in the primary MINVI trial (NCT03631940) will collect Near Infrared Spectroscopy (NIRS) data in the first 10 minutes of life on a subset of 200 non-vigorous term and near-term infants enrolled in the trial.

DETAILED DESCRIPTION:
Rationale: Caregivers and researchers raised theoretical concerns that the UCM technique may deliver blood rapidly toward a non-vigorous newborn predisposing them to higher rates of brain injury or dislodging cellular debris into the brain. However, of the 13 studies on term infants comparing UCM to ECC, none have reported adverse outcomes. Even in more fragile preterm infants, no harm has been reported. All demonstrated improvements similar to DCC with increased red cell mass (measured by hematocrit or hemoglobin) improved blood pressure, increased pulmonary blood flow and improved ferritin at 6 weeks to 6 months of age with UCM. Nevertheless, careful assessment of safety is essential. Immediate physiological measurements on a subset (n=200) of infants of the two sub-study sites where the use of NIRS is standard of care, University of Alberta and SMBHWN, to establish the safety and efficacy of UCM. This aim will further test our hypotheses that infants in the UCM group will have improved early cardiac and cerebral hemodynamics within the first 10 minutes.

The Near-infrared spectroscopy (NIRS) is a technology that allows non-invasive continuous real-time measurement of the regional tissue oxygen saturation (StO2) of organs such as the brain. There are well-established reference cerebral StO2 values for uncomplicated term and preterm deliveries; however, there are no completed RCTs using NIRS in the delivery room. Our group is currently leading the first multicenter trial (1R01HD088646-01A1) comparing DCC and UCM measuring NIRS at birth in premature infants. If cerebral oxygenation is improved, it will provide one plausible explanation for the long-term benefits expected with UCM. While published data exists on cerebral oxygenation directly comparing UCM with DCC, some studies demonstrated increases in cerebral oxygenation at 4 hours of age with DCC, and a decrease in cerebral oxygenation at birth with DCC compared to immediate cord clamping. To our knowledge, no studies using cerebral oxygenation in non-vigorous term/near-term infants have ever been performed. This sub-study (n=200) will yield the largest available sample of specific measurements of cerebral oximetry in non-vigorous term newborns.

Substudy Sites: Three sites experienced with NIRS (University of Alberta, Sharp Grossmont Hospital and SMBHWN) will obtain and report the physiological changes with UCM and ECC at 10 minutes of life. Data from the non-invasive monitoring devices are recorded using a continuous real-time data acquisition system that provides a second-by-second record of the resuscitation that is also time-linked to the video recordings. Both sites have 24/7 research team coverage that attend all high-risk deliveries. The research team will ensure accurate sensor placement and data collection. These two exceptional settings will allow us to collect significant data regarding resuscitation outcomes linked to cerebral oxygenation.

Protocol for NIRS Sub-Study: At the two sub-study sites, the use of NIRS is standard of care.

As part of the NIRS sub-study, sites will collect physiological and resuscitation data from birth (mean airway pressure, fractional oxygen) in addition to cerebral oxygenation. Once the newborn is delivered, receives the intervention (UCM or ECC), and is stabilized during resuscitation, a NIRS sensor (Fore-Sight, CAS Medical, Branford, CT) will be placed on the right forehead within 10 minutes of the newborn being placed on the warmer. While arterial saturation and heart rate data will be available to the clinical team, data from NIRS will be blinded. Data on all study infants will be recorded for the first 10 minutes in the delivery room at the two sites. Heart rate, oxygen saturations, and cerebral oxygenation will be downloaded as per both site's practice for neonatal resuscitation.

ELIGIBILITY:
Inclusion Criteria:

* Non-vigorous newborns born between 35-42 weeks gestation
* Born at NIRS Sub-study site

Exclusion Criteria:

* Known major congenital or chromosomal anomalies of newborn
* Known cardiac defects other than small ASD, VSD and PDA
* Complete placental abruption/cutting through the placenta at time of delivery
* Monochorionic multiples
* Cord Avulsion
* Presence of non-reducible nuchal cord
* Perinatal providers unaware of the protocol
* Incomplete delivery data Infants born in extremis, for whom additional treatment will not be offered

Ages: 35 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2022-12-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anup Katheria, MD, Principal Investigator — Sharp Mary Birch Hospital for Women & Newborns
Locations (3):
- United States (2):
  - Sharp Grossmont Hospial, San Diego, California
  - Sharp Mary Birch Hospital for Women and Newborns, San Diego, California
- Governors of University of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Katheria AC, Law BHY, Poeltler D, Rich W, Ines F, Schmolzer GM, Lakshminrusimha S. Cardiac and cerebral hemodynamics with umbilical cord milking compared with early cord clamping: A randomized cluster crossover trial. Early Hum Dev. 2023 Mar;177-178:105728. doi: 10.1016/j.earlhumdev.2023.105728. Epub 2023 Feb 14. PMID 36827750

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Umbilical Cord Milking | Early Cord Clamping
Started | 15 | 19
Completed | 15 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Umbilical Cord Milking | Early Cord Clamping | Total
Number analyzed (Participants) | 15 | 19 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 19 | 34
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Gestational Age in weeks] | 38.13 (1.56) | 38.95 (1.72) | 38.54 (0.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 16
  Male | 9 | 9 | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 10 | 0 | 10
  United States | 5 | 19 | 24

OUTCOME MEASURES:

1. Primary Outcome: StO2 in the First 10 Minutes of Life
Description: Cerebral oxygenation derived from skeletal muscle oxygen saturation (StO2) measured by near-infrared spectroscopy (NIRS). Once the newborn is delivered, receives the intervention (UCM or ECC), and is stabilized during resuscitation, a NIRS sensor (Fore-Sight, CAS Medical, Branford, CT) will be placed on the right forehead within 10 minutes of the newborn being placed on the resuscitation bed.
Time Frame: birth to 10 minutes of life
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Umbilical Cord Milking | Early Cord Clamping
Number analyzed (Participants) | 15 | 19
percent | 70 (7.15) | 74.5 (2.17)

2. Secondary Outcome: Heart Rate at 10 Minutes
Description: Heart rate was recorded from the electrocardiogram monitor.
Time Frame: Birth to 10 minutes of life
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Umbilical Cord Milking | Early Cord Clamping
Number analyzed (Participants) | 15 | 19
Beats per minute | 152 (12.76) | 160 (12.99)

ADVERSE EVENTS:
Time Frame: The first 10 minutes of life.
Arm/Group | Umbilical Cord Milking | Early Cord Clamping
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/19
Other Adverse Events (participants affected / at risk) | 0/15 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2022-11-16): https://cdn.clinicaltrials.gov/large-docs/56/NCT03621956/Prot_000.pdf